CLINICAL TRIAL: NCT00708032
Title: Clinical Performance of a New Daily Disposable Contact Lens Worn in a Neophyte Population.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0806
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Refractive Error; Myopia
MeSH Terms: conditions — Refractive Errors; Myopia | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- spectacles (Other): habitual spectacles worn daily for 12 months
  Interventions: Device: spectacles
- narafilcon A soft contact lenses (Experimental): narafilcon A soft contact lenses worn as daily disposable for 12 months
  Interventions: Device: narafilcon A soft contact lenses

INTERVENTIONS:
Device: spectacles — habitual spectacles
  Arms: spectacles
Device: narafilcon A soft contact lenses — narafilcon A daily disposable contact lenses
  Arms: narafilcon A soft contact lenses

SUMMARY:
This study seeks to evaluate the impact of wearing a new daily disposable soft contact lens on the neophyte population.

ELIGIBILITY:
Inclusion Criteria:

1. They are of legal age (18 years) and capacity to volunteer.
2. They understand their rights as a research subject and are willing to sign a Statement of Informed Consent.
3. They are willing and able to follow the protocol.
4. They would be expected to attain at least 6/9 (20/30) in each eye with the study lenses.
5. They are able to wear contact lenses with a back vertex power of -1.00 to -6.00DS.
6. They have a maximum of 1.00D of refractive astigmatism (i.e. ≤ 1.00 DC).
7. They have successfully worn contact lenses within six months of starting the study.

Exclusion Criteria:

1. They have an ocular disorder which would normally contra-indicate contact lens wear.
2. They have a systemic disorder which would normally contra-indicate contact lens wear.
3. They are using any topical medication such as eye drops or ointment.
4. They are aphakic.
5. They have had corneal refractive surgery.
6. They have any corneal distortion resulting from previous hard or rigid lens wear or has keratoconus.
7. They are pregnant or lactating.
8. They have grade 2 or greater of any of the following ocular surface signs: corneal oedema, corneal vascularisation, corneal staining, tarsal conjunctival changes or any other abnormality which would normally contraindicate contact lens wear.
9. They have any infectious disease (e.g. hepatitis) or any immunosuppressive disease (e.g. HIV).
10. They have diabetes.
11. They have taken part in any other clinical trial or research, within two weeks prior to starting this study.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2008-06-01 (Actual); Primary Completion 2009-12-01 (Actual); Study Completion 2009-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eurolens Research, The University of Manchester, Manchester, Greater Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 74 subjects enrolled into the study, 38 into the TruEye group and 36 in the spectacle group. Forty-eight subjects completed the study.
Groups:
- Spectacles: spectacles worn daily for 12 months
- Narafilcon A Lenses: narafilcon A soft contact lenses worn as daily disposable for 12 months
Period: Overall Study
Arm/Group | Spectacles | Narafilcon A Lenses
Started | 36 | 38
Completed | 26 | 22
Not Completed | 10 | 16
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Pregnancy | 0 | 1
Not completed — Poor vision | 0 | 6
Not completed — Visit out of range at month 12 | 4 | 1
Not completed — Did not meet protocol criteria | 1 | 2
Not completed — Protocol Violation | 4 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: There were 74 subjects enrolled with 48 completing the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Spectacles | Narafilcon A Lenses | Total
Number analyzed (Participants) | 36 | 38 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (8.1) | 26.5 (7.4) | 26.5 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 20 | 19 | 39
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 36 | 38 | 74

OUTCOME MEASURES:

1. Secondary Outcome: Biomicroscopy Findings After 12 Months of Daily Wear From Slit Lamp Analysis.
Description: Comprised of 8 categories (conjunctival hyperemia, limbal hyperemia, corneal vascularization, microcysts, Oedema, corneal staining, conjunctival staining and papillary conjunctivitis) each scored on a scale of 0 to 4 where 0=none, and 4=maximum score for each category.
Time Frame: at 12 months
Population: Subjects analyzed were those who were enrolled, randomized to a study arm, and completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Narafilcon A Lenses | Spectacles
Number analyzed (Participants) | 22 | 26
units on a scale
  Conjunctival Hyperemia | 1.09 (0.22) | 1.00 (0.22)
  Limbal Hyperemia | 0.89 (0.25) | 0.80 (0.24)
  Corneal Vascularization | 0.00 (0.00) | 0.00 (0.00)
  Microcysts | 0.00 (0.00) | 0.00 (0.00)
  Oedema | 0.00 (0.00) | 0.00 (0.00)
  Corneal Staining | 0.33 (0.32) | 0.25 (0.27)
  Conjunctival Staining | 0.83 (0.40) | 0.22 (0.15)

2. Secondary Outcome: Visual Acuity After 12 Months of Wear
Description: Visual acuity is measured at high and low contrasts, via the Snellen scale which is then mathematically converted to logMar units. High contrast refers to a darker print on the Snellen chart and is an easier testing environment compared to the low contrast which has a grayer print.
Time Frame: at 12 months
Population: Subjects analyzed were those who were enrolled, randomized to a study arm, and completed the study.
Measure: Mean (Standard Deviation); unit: logMar
Arm/Group | Narafilcon A Lenses | Spectacles
Number analyzed (Participants) | 22 | 26
logMar
  High Contrast | -0.05 (0.08) | -0.11 (0.06)
  Low Contrast | 0.29 (0.11) | 0.18 (0.07)

3. Secondary Outcome: Subjective Overall Comfort After 12 Months of Daily Wear
Description: subject response using a scale of 0 to 100, where 0 = poor comfort, 100 = excellent comfort
Time Frame: at 12 months
Population: Subjects analyzed were those who were enrolled, randomized to a study arm, and completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Narafilcon A Lenses | Spectacles
Number analyzed (Participants) | 22 | 26
units on a scale | 87.8 (10.0) | 82.2 (15.1)

4. Secondary Outcome: Subjective Overall Vision After 12 Months of Daily Wear
Description: subject response using a scale of 0 to 100, where 0 = poor vision, 100 = excellent vision
Time Frame: at 12 months
Population: Subjects analyzed were those who were enrolled, randomized to a study arm, and completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Narafilcon A Lenses | Spectacles
Number analyzed (Participants) | 22 | 26
units on a scale | 88.7 (11.5) | 82.5 (15.1)

5. Primary Outcome: Papillary Conjunctivitis
Description: Papillary conjunctivitis which is collected as part of the biomicroscopy data and is identified from a slit lamp examination. Grade 0 to Grade 4 with grade 0 implying no health concerns.
Time Frame: 12 months
Population: Subjects analyzed were those who were enrolled, randomized to a study arm, and completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Narafilcon A Lenses | Spectacles
Number analyzed (Participants) | 22 | 26
units on a scale | 1.22 (0.21) | 1.04 (0.26)

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the sutdy. Approximately 12 month.
Arm/Group | Spectacles | Narafilcon A Lenses
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/38
Other Adverse Events (participants affected / at risk) | 5/36 | 4/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spectacles (N=36) | Narafilcon A Lenses (N=38)
Non-signficant Corneal Event (Eye disorders) | 5 (27) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication requires agreement and written consent from the Sponsor.